CLINICAL TRIAL: NCT05821244
Title: Feasibility of Manipulating Exercise Timing in Breast Cancer Survivors on Chemotherapy
Brief Title: Exercise Timing in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adriana Coletta, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00162526
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Exercise; Resistance Training; Aerobic Exercise; Exercise Time-of-Day; Breast Cancer; Breast Cancer Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Group (Experimental): Participants must start their exercise between the hours of 5am and 10am.
  Interventions: Behavioral: Exercise Timing Groups
- Evening Group (Experimental): Participants must start their exercise between the hours of 3pm and 8pm.
  Interventions: Behavioral: Exercise Timing Groups

INTERVENTIONS:
Behavioral: Exercise Timing Groups — Individualized resistance training program, consisting of twice weekly training sessions supervised via telehealth with a cancer exercise trainer.

SUMMARY:
The purpose of this study is to demonstrate the feasibility of assigning breast cancer survivors currently receiving chemotherapy to exercise at a specific time of day, e.g., morning or afternoon/evening, for a 4-week exercise intervention. Information gathered from this study will help inform a future, larger trial.

Study Aims:

1. Assess the feasibility of engaging in exercise at an assigned time-of-day (e.g., morning or afternoon/evening) in breast cancer survivors on chemotherapy. Hypothesis: Assigning windows of time within the day to complete exercise (e.g. 5-10am exercise start time vs. 3-8pm exercise start time) will be feasible among this patient population.

1a. Determine the acceptability engaging in exercise at an assigned time-of-day (e.g., morning or afternoon/evening) in breast cancer survivors on chemotherapy. Hypothesis: Engaging in exercise at an assigned time-of-day will be acceptable in this patient population.

2. To generate evidence on the magnitude of the effect sizes and outcome variability of physical function and human performance variables. Tests to be conducted at baseline and end of study to measure physical function and human performance variables include: Timed up and go test, 30-second chair stand, handgrip strength, cardiorespiratory fitness.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to an exercise timing group (AM or PM), of which they will be required to complete their exercise during a specific time of day. Participants randomized to the AM group will be required to start their exercise between 5am and 10am for the duration of the 4-week intervention. Participants randomized to the PM group will be required to start their exercise between 3pm and 8pm.

At baseline and end of study assessments, participants will complete the following physical tests to evaluate physical function, strength, and cardiorespiratory fitness: timed up and go test, 30-second chair stand test, handgrip strength test, cardiorespiratory fitness test. These tests and assessments will be carried out with the Huntsman Cancer Institute (HCI) Wellness Center's Personal Optimism With Exercise Recovery (POWER) program. These tests will occur at the HCI Wellness Center gym. At the end of study assessments participants will also be asked to complete an exit survey, and two short questionnaires related to sleeping and eating habits.

Participants will complete two personalized resistance exercise training sessions supervised by a Cancer Exercise Specialist via the telehealth platform in the electronic medical record. These resistance training sessions are part of the POWER program. Participants will also be required to engage in weekly, moderate-intensity aerobic exercise, with the goal of completing 90 minutes of aerobic exercise per week. The type of aerobic exercise engaged in (e.g., walking, biking, hiking, etc), and location to complete the aerobic exercise (e.g., at home, local park, local gym, HCI Wellness Center gym, etc.) is the participant's choice. Participant's will be required to submit weekly aerobic exercise training logs.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III Breast Cancer patients with plans to start chemotherapy or just started chemotherapy. Just started chemotherapy is defined as already receiving one cycle of chemotherapy.
* ECOG 0, 1, 2

Exclusion Criteria:

* Stage IV Breast cancer patients
* ECOG >/= 3
* Stage I-III Breast Cancer patients who do not have plans to start chemotherapy or who have received more than one cycle of breast cancer chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | through study completion, on average four weeks
  The proportion of patients who complete at least 75% of their assigned workouts within the time-of-day window assigned throughout the four-week assessment period

SECONDARY OUTCOMES:
Acceptability | through study completion, on average four weeks
  Study acceptability will be measured as the proportion of patients who qualitatively report a positive response to at least half of exit survey themes.
Whole body physical function | Baseline and through study completion, on average four weeks
  Timed up and go test
Lower body physical function | Baseline and through study completion, on average four weeks
  30-second chair stand test
Whole body strength | Baseline and through study completion, on average four weeks
  Handgrip strength test
Cardiorespiratory fitness | Baseline and through study completion, on average four weeks
  Cardiorespiratory fitness test

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Coletta, PhD, MS, RD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available